CLINICAL TRIAL: NCT00224887
Title: Family-Based Nutrition Intervention for Latino Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 320; R01HL070218 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Heart Diseases
MeSH Terms: conditions — Obesity; Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- in home nutrition counseling (Experimental): In-home family-based behavioral counseling using in-person and video interventions delivered by community health advisors
  Interventions: Behavioral: In home nutrition counseling
- standard nutrition education curriculum (Active Comparator): standard nutrition education curriculum consisting of video and lesson plans based on USDA Food Guide pyramid
  Interventions: Other: standard nutrition education curriculum

INTERVENTIONS:
Behavioral: In home nutrition counseling — In home family-based behavioral counseling
  Arms: in home nutrition counseling
Other: standard nutrition education curriculum — video and lesson plans based on USDA Food Guide Pyramid
  Arms: standard nutrition education curriculum

SUMMARY:
Primary Hypothesis Children whose mothers receive the FBC sessions will have significantly lower BMI one year after the intervention compared to control group children whose families receive an active placebo control.

Secondary Hypotheses In families that receive the FBC, household availability of fruits and vegetables will increase, and availability of high fat foods will decrease, as measured by multiple household food inventories, compared to control group families exposed to an active placebo intervention.

Household level of food security, mothers' food purchase motives and family food interaction will influence the effects of the FBC on household food supplies.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease accounted for 40.6% of deaths in the United States in 1998. Although CVD does not manifest until adulthood, risk factors for CVD, such as obesity, may develop in childhood and persist into adulthood. We propose to test the efficacy of an intervention designed to prevent obesity in low-income, Mexican American children. Mexican-American children are more obese than other minority groups in the U.S. population, and are the fastest growing minority group in the U.S.A. Poor dietary practices, especially food habits that are acquired as families acculturate to the American food supply, are thought to be associated with children's excess weight gain.

We propose to conduct a randomized clinical trial in which 150 families receive family-based behavioral counseling (FBC) sessions and 150 families receive an active placebo control intervention. Mothers and their second or third grade children from sixteen low-wealth elementary schools will be randomized into either the treatment or control interventions. The purpose of the FBC sessions is to change children's food environment. Specifically, we intend to increase the amount of fruit and vegetables, and decrease the amount of high fat foods available to children in their homes. In addition, we will encourage parents to model healthy dietary practices for their children. Two intervention strategies, a video, "What's to Eat?" developed for this population and photographs of each family's food practices, taken by family members, will be used in the counseling sessions. The control intervention will consist of group sessions using a curriculum that adapts standard nutrition recommendations for traditional Mexican-American foods. Community health advisors will conduct both the FBC and control sessions. The primary outcome of the trial is children's BMI. The secondary outcome is household food supplies. We hypothesize that within a one year timeframe, children's whose mothers are exposed to the FBC will have lower BMI's compared to children whose mothers receive the active placebo control intervention. The mechanism through which we intend to change weight status is altering the type of foods available to children in their homes. Therefore, two household food inventories, one collected prior to and one after the family's payday will be used as secondary outcomes. In addition, mothers' reports of household food security level, food purchase motives, and family food interaction will be collected as covariates. Measurements will be collected within one month of completing the interventions and at six months and one year follow-up.

DESIGN NARRATIVE:

Family Based Counseling. Community health advisors visit mothers who are randomly assigned to the FBC sessions once a month, for six months, in their homes. During the first session, mothers watch the video, "What's to Eat?" with the CHA and discuss food related parenting issues. In the subsequent five sessions, photographs of the family's food habits, taken by mothers, are used as visual aids for the intervention sessions. In addition, at each session, the CHA provides mothers with a food sample related to their dietary change goal. Examples of the types of foods provided to families include fat free milk, cooking oil spray, fruits and vegetables or low fat yogurt.

Group Based Nutrition Sessions Families assigned to the group sessions are invited to one group session a month for six months. Group sessions are held in the morning and the evening to accommodate mothers' schedules. The groups sessions are based on a standard Mexican-American nutrition curriculum. This curriculum consists of a video and five lesson plans based on the USDA Food Guide Pyramid that emphasize foods indigenous to the Mexican diet. In addition to lessons from the curriculum, nutrition games, based on popular game shows such as "Nutrition Jeopardy" and "Family Feud" are also played during the sessions.

Primary Outcome Measure - Children's Weight Status Height & Weight: Standing height will be measured twice, to the nearest millimeter, using a portable direct reading stadiometer. If the two measures differ by more than 5 mm, a third measure will be obtained. Body weight will be measured twice, to the nearest 0.1 kg, using digital scales with subjects wearing light indoor clothing without shoes. If the two measures differ by more than 0.2 kg, a third measure will be obtained. The mean of the two measures, or the median of three measures, are used to calculate BMI.

Secondary Outcome Variable Our intervention is designed to prevent obesity in children by changing their food environments. Therefore, the secondary outcome for this research is changes in the type of food available to children in their homes. Specifically, a, quantitative household food inventory that assess the actual amount of fruit, vegetables, high fat foods and total food energy is collected. Inventories are collected within three days of grocery shopping. Two trained research assistants conduct each inventory, which require approximately 15 to 60 minutes to complete. All foods except spices, hot sauces, baking powder, baking soda, coffee, tea and spoiled foods are collected in the inventories. The amounts listed on the label of packaged, canned, or frozen foods are recorded, and if opened, the proportion remaining in the package is recorded. The amount of meat or cheese is recorded in pounds based on the package label. The number of fresh fruits, vegetables and eggs are counted. Beverages are recorded in fluid ounces or gallons. Prepared foods on the stove or leftover in the refrigerator are estimated in cups.

Mothers' Socio-environment Measurements Demographics: Demographic variables, including household composition, who in the household shares the same food supplies, and where mothers purchase or receive food supplies (including WIC or food donations) will be collected from the mothers. To examine the variability in household food supplies relative to pay day, mothers will also report when their family receives pay checks. Children's demographic variables will include gender, age, and grade level.

Household Level of Food Security: Food security is defined as people's assured access to enough acceptable food, that is acquired in socially acceptable ways, for an active and healthy life. This construct will be measured using the 18 item U.S.D.A. Core Food Security Module (FSM). This instrument conceptualizes food security as consisting of four components: 1) quantity of food, 2) quality of food, 3) food anxiety and 4) food acquisition in socially acceptable ways (166, 167). Households are categorized into four levels of food insecurity: 1) food secure, 2) food insecure without hunger, 3) food insecure with moderate hunger and 4) food insecure with severe hunger (i.e., children's food intake is restricted).

ELIGIBILITY:
The inclusion criteria for the study are:

1. Ethnicity: Mother is of Mexican descent and identifies with the Mexican-American community.
2. Age: Child is between 6 and 9 years 11.9 months old.
3. Family lives in the San Jose area
4. Family does not plan to move out of the area within the next 12 months.

The exclusion criteria for the study are:

1. Metabolic disease/syndrome associated with obesity.
2. Diabetes
3. Chronic gastro-intestinal disease
4. Chronic renal disease
5. Heart disease
6. Eating disorders
7. Aids/HIV infection
8. Use of steroids
9. Use of insulin injections
10. Use of oral antidiabetic agents
11. Use of thyroid hormones
12. Use of growth hormones
13. Other diseases or use of other medications that may impact growth based on Dr. Mendoza's assessment.
14. Family shares food with 2 other families with children under the age of 12.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

IPD SHARING:
Plan to Share IPD: No
No plan to share data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | in Home Nutrition Counseling | Standard Nutrition Education Curriculum
Started | 154 | 153
Completed | 148 | 147
Not Completed | 6 | 6
Not completed — Pregnancy | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | in Home Nutrition Counseling | Standard Nutrition Education Curriculum | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (1.2) | 7.8 (1.1) | 7.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 104 | 221
  Male | 37 | 49 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Body Mass Index (BMI)
Description: child's Body Mass Index
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | in Home Nutrition Counseling | Standard Nutrition Education Curriculum
Number analyzed (Participants) | 154 | 153
kg/m^2 | 0.52 (1.56) | 0.66 (1.43)

ADVERSE EVENTS:
Time Frame: 12 months
Description: The study was considered to be minimal risk. Interventions were informational/educational and did not include medications or invasive testing/procedures.
Arm/Group | in Home Nutrition Counseling | Standard Nutrition Education Curriculum
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/153
Other Adverse Events (participants affected / at risk) | 0/154 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes